CLINICAL TRIAL: NCT00533598
Title: A Study to Determine the Effects of MK0557 in Obese Subjects (0557-006)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0557-006; 2007_613
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — spiro(cyclohexane-1,3'(1'H)-furo(3,4-C)pyridine)-4-carboxamide, N-(1-(2-fluorophenyl)-1h-pyrazol-3-yl)-1'-oxo-, trans-

INTERVENTIONS:
Drug: MK0557

SUMMARY:
The purpose of this study is to assess the effects of MK0557 on body weight in obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 21 and 65 years of age, willing to avoid all prescription and nonprescription medicine to alter body weight for entire study

Exclusion Criteria:

* You are or plan to become pregnant
* You have smoked or used nicotine within 6 months of the study
* History of abusing alcohol and/or drugs
* History of a stroke, you have diabetes mellitus, you are taking medication for high blood pressure, you have had recent surgery, you have been involved in another study within 3 months of study, use of cholesterol or anti-seizure medication during the study
* Have participated in a weight loss program 3 months before the study or during the course of the study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-09; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC